CLINICAL TRIAL: NCT01456806
Title: Programme of Diabetes Education in the City of Corrientes (PRODIACOR): Clinical, Metabolic and Economic Outcomes of a Prospective-randomized Trial Based on Different Patient-centered Educational Strategies for People With Type 2 Diabetes
Brief Title: Educative Intervention to Improve Type 2 Diabetes Mellitus Control in Corrientes
Acronym: PRODIACOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Endocrinologia Experimental y Aplicada (Other)
Collaborators: National Council of Scientific and Technical Research, Argentina (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: 1374/2006 (ACC)
Record Dates: First submitted 2011-10-19; First posted 2011-10-21 (Estimated); Last update posted 2011-10-21 (Estimated); Status verified 2011-10

CONDITIONS: Type 2 Diabetes
Keywords: T2DM; Cardiovascular risk factors; Metabolic control; Well-being; Cost; Cost-consequence
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Patients and provider non educated (No Intervention): In this arm neither the patients nor the providers have attended the groupal education courses
  Interventions: Other: Education
- Provider educated (Active Comparator): Provider attend the interactive group education, while patients do not.
  Interventions: Other: Education
- Patients Educated (Active Comparator): Patients attend the interactive group education, while providers do not.
  Interventions: Other: Education
- Providers/Patients Educated (Active Comparator): Provider and Patients both attend the interactive group education.
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — Structured group education programmes were delivered to provider and/or people with type 2 diabetes by trained professionals; identical system interventions were applied to all four groups.
  Other Names: Diabetes Education

SUMMARY:
Objective: To evaluate the effect of system interventions (data recording procedures and complete coverage of medications and supplies) with or without physician and/or patient education, upon the psychological, clinical, metabolic and therapeutic indicators and the costs of care of people with type 2 diabetes.

Design: Randomized 2x2 design; sample size was determined considering the change in haemoglobin A1c (primary outcome variable) using a two-sided test at the 5% level of significance, and 80% power using a paired t-test. Sample size was increased by 25% to account for non-independence and patient drop-out.

Setting: Primary care level in the city of Corrientes, Argentina with involvement of all three Argentinean health subsectors (public health, social security and the private, prepaid system).

Participants: 36 general practitioners and 468 adults (62-71% women, mean age 62 years) with type 2 diabetes. Patients of the participating physicians (nine in each group), were randomly selected and assigned to one of four groups (117 patients each): control, provider education, patient education, and provider/patient education.

Intervention: Structured group education programmes were delivered to provider and/or people with type 2 diabetes by trained professionals; identical system interventions were applied to all four groups.

Main outcome measures: Body mass index, blood pressure, fasting glucose, haemoglobin A1c levels, lipid profile, drug consumption, resource use, and patient well being (WHO-5 questionnaire and Lowe score), at baseline and up to 42 months at every 6 months intervals.

DETAILED DESCRIPTION:
The study protocol was evaluated and approved by an external ethical committee; patients gave informed consent to participate in the study according with the guidelines from the International Conference on Harmonisation and WHO good clinical practice standards. The study design has been previously described in detail.30 Briefly, the investigators implemented a randomized 2x2 design to address the effectiveness of different education strategies involving the health provider and people with diabetes).

Sample size: for its determination in each of the four groups, the investigators considered the change in haemoglobin A1c (from baseline to the end of the study) as the primary outcome variable. This was done using a two-sided test at the 5% level of significance and 80% power using a paired t-test. The sample size was increased by 25% to account for non-independence and dropout, resulting in the number of providers and patients listed in table 1.

Educational strategies The investigators used the Diabetes Training Course for Physicians and Diabetes Structured Education Courses for People with T2DM, whose characteristics and usefulness have been previously reported.

Data collection Patients' clinical, psychological, biochemical, therapeutic and economic data before and after PRODIACOR were recorded using the Physician Data Form, the Annual and Bi-annual Clinical Record Form and the Feedback Report Form. The investigators developed software that compares the first two mentioned forms and generates a Biannual Feedback Report for physicians and patients; it compares the values recorded for haemoglobin A1c, serum lipids and blood pressure, and the goal proposed for each parameter according to international standards. It also includes recommendations about appropriate treatment to achieve therapeutic goals.31 Additionally, the investigators used the Patient Questionnaire, based on the one previously used in the Diabetes Advantage Program (DAP) which includes questions about the disease, and the WHO-5 well-being questionnaire. Data collection was completed with the Personalized Checkbook, a tool initially developed for the PROPAT study, whose aim and content have been previously described. It serves to order procedures, consultations, laboratory tests, prescription of drugs and strips for glucose self-monitoring, to record and communicate results, and as a payment voucher for all those items.

Study and Data management The Local Coordinator (city of Corrientes) together with the Central Cordinating Center (CENEXA), oversaw the education courses and the overall trial and maintained periodic contact with the participating physicians. Performance of the physicians and their patients was monitored at regular intervals (6 months) during the whole study period. Every physician was visited twice a year by a physician monitor who assessed the quality of the data he has recorded.30 Participating physicians collect their own patients´ data, sent it to the Local Coordinator who controlled its completeness and forwarded to the Central Coordinating Centre.

Resource utilization and costs The data recorded include all direct medical items used by each of the patients ascribed to the programme, and were obtained from the checkbook and the utilization and cost records from each of the participating health coverage entities.

Utilization was classified into five groups: i) hospitalizations, ii) drugs and supplies, iii) diagnostic tests, iv) special studies, and v) physician office visits. Drugs were identified by their generic and commercial name and their corresponding presentation. Their costs were assessed from retail prices published by Alfabeta.net and adjusted to July 2004 using the health chapter of local Consumer Price Index.

Estimated drug costs and haemoglobin A1c reduction experienced by each treatment group were used to construct marginal figures of cost-consequence ratio. For this purpose, the investigators calculated such ratio figures for each experimental group, i.e., the investigators expressed the total drug cost associated to 1% haemoglobin A1c decrease to 10 mm Hg of systolic blood pressure or 10 mg/dL of triglyceride levels. The investigators did not currently estimate the costs of the educational interventions themselves, namely, all the physical and human resources involved in the management and administrative activities of the programme.

Statistical analysis To estimate the effects of the different educational interventions tested, intention to treat analysis was used. Initial univariate differences among groups for quantitative data were analyzed by one-way ANOVA (Bonferroni post hoc test). Factorial ANOVA and two-way ANOVA models (Bonferroni post hoc test) were used to assess the differences among groups along the study. ANOVA was also used to explore initial vs. end-of-study differences among quantitative data. Differences among qualitative measures were explored by Chi-squared (Yates corrected). P values of less than 0.05 were considered as significant (two tailed). Missing data strategies applied to the primary endpoint were last observation carried forward and complete case analysis. Both strategies were compared to evaluate the impact of missing data on the efficacy analysis of the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Adults Patients with type 2 diabetes
* Being regularly attended at the doctors office during at least one year

Exclusion Criteria:

* Newly diagnosed type 2 diabetes
* Advanced stage of chronics complications (End-stage-kidney disease)
* Heart Failure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2006-12; Primary Completion 2007-03 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
HbA1c | 42 months

SECONDARY OUTCOMES:
Quality of Care Indicators | 42 months
  Body mass index, blood pressure, fasting glucose, lipid profile, drug consumption, resource use, and patient well being (WHO-5 questionnaire and Lowe score)

CONTACTS AND LOCATIONS:
Overall Officials: Juan J Gagliardino, MD, Study Director — CENEXA (UNLP-CONICET La Plata)
Locations (1):
- CENEXA (UNLP-CONICET La PLata), La Plata, Buenos Aires, Argentina

REFERENCES:
- [Background] Gagliardino JJ, Lapertosa S, Villagra M, Caporale JE, Oliver P, Gonzalez C, Siri F, Clark Ch Jr; PRODIACOR. PRODIACOR: a patient-centered treatment program for type 2 diabetes and associated cardiovascular risk factors in the city of Corrientes, Argentina: study design and baseline data. Contemp Clin Trials. 2007 Jul;28(4):548-56. doi: 10.1016/j.cct.2007.01.004. Epub 2007 Jan 12. PMID 17331807
- [Derived] Gagliardino JJ, Lapertosa S, Pfirter G, Villagra M, Caporale JE, Gonzalez CD, Elgart J, Gonzalez L, Cernadas C, Rucci E, Clark C Jr; PRODIACOR. Clinical, metabolic and psychological outcomes and treatment costs of a prospective randomized trial based on different educational strategies to improve diabetes care (PRODIACOR). Diabet Med. 2013 Sep;30(9):1102-11. doi: 10.1111/dme.12230. Epub 2013 Jun 7. PMID 23668772